CLINICAL TRIAL: NCT04474899
Title: Sympathoinhibition as a Preferred Second Line Treatment of Obesity Related Hypertension
Acronym: OHT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Perth Hospital (Other)
Collaborators: The University of Western Australia (Other)
Responsible Party: Principal Investigator, Dr Markus Schlaich, Principal Investigator, Royal Perth Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-4-1-7565
Record Dates: First submitted 2020-06-03; First posted 2020-07-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — moxonidine; Amlodipine

STUDY DESIGN:
Intervention Model Description: Randomized, double blind cross over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Experimental): Moxonidine 0.4mg/daily
  Interventions: Drug: Moxonidine 0.4 MG; Drug: Amlodipine 5mg
- Phase 2 (Experimental): Amlodipine 5mg
  Interventions: Drug: Moxonidine 0.4 MG; Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: Moxonidine 0.4 MG — Participants will be randomly assigned to receive moxonidine 0.4mg/daily and will later receive the alternate treatment. As the study is double blind neither the participant nor the study personnel will be aware of which treatment is currently being tested to avoid any effect this may have on the results. The two 12-week treatment phases will be separated by a 6-week wash out (drug-free) period.
Drug: Amlodipine 5mg — Participants will be randomly assigned to receive amlodipine 5mg and will later receive the alternate treatment. As the study is double blind neither the participant nor the study personnel will be aware of which treatment is currently being tested to avoid any effect this may have on the results. The two 12-week treatment phases will be separated by a 6-week wash out (drug-free) period.

SUMMARY:
This study is designed to investigate whether sympathoinhibition with moxonidine could provide added metabolic benefit compared to the second line therapy in the current guidelines.

DETAILED DESCRIPTION:
This is a randomised, double-blind, cross-over study. Participants will be randomly assigned to receive either moxonidine 0.4mg daily or amlodipine 5mg and will later receive the alternate treatment.

Comprehensive testing will occur after each 12 week treatment phase and will include assessment of muscle sympathetic nerve activity, gut microbiome analysis and metabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 -70 years
* (Body Mass Index) BMI≥30kg/m2
* Currently weight stable (+/- 3% in previous 6-12 months and not on any specific exercise or dietary program)
* Elevated clinic systolic (Blood Pressure) BP ≥135 or diastolic BP ≥85mmHg,
* on ACE inhibitor for at least 6 weeks prior to baseline assessment

Exclusion Criteria:

* Grade 2-3 hypertension (systolic office BP >160, diastolic office BP >100 mmHg)
* Secondary causes of hypertension
* CKD (Chronic kidney disease) stage 4-5 {(estimated glomerular filtration) eGFR<30ml/min}
* Heart failure NYHA (New York Heart Association) class II-IV
* Recent CV (cardiovascular) event (acute myocardial infarction, acute coronary syndrome, stroke or transient ischaemic attack within the previous six months) unstable psychiatric condition
* medication such as corticosteroids, several antidepressants and antipsychotics
* Female participants of childbearing potential must have a negative pregnancy test prior to treatment

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06-24 (Actual); Primary Completion 2024-02-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 30 weeks
  Both Systolic and diastolic blood pressure assessed by office and ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
blood glucose levels | 30 weeks
  Changes in glycemic control through oral glucose tolerance test
Gut microbiota profile | 30 weeks
  Change in gut microbiota assessed by short chain fatty acid
Lipid levels in blood | 30 weeks
  change in triglyceride, HDL and LDL levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD, Principal Investigator — University of Western Australia and Royal Perth Hospital
Locations (1):
- Dobney Hypertension Centre, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared to maintain anonymity and confidentiality of the participants

REFERENCES:
- [Background] Carnagarin R, Gregory C, Azzam O, Hillis GS, Schultz C, Watts GF, Bell D, Matthews V, Schlaich MP. The Role of Sympatho-Inhibition in Combination Treatment of Obesity-Related Hypertension. Curr Hypertens Rep. 2017 Oct 28;19(12):99. doi: 10.1007/s11906-017-0795-1. PMID 29080925